CLINICAL TRIAL: NCT04811638
Title: The Validity and Reliability of the Turkish Version of the Chelsea Critical Care Physical Assesment Tool
Brief Title: The Validity and Reliability Study of the Chelsea Critical Care Physical Assesment Tool
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Medical Park Hospital Istanbul (Other)
Responsible Party: Principal Investigator, Mehmet Burak Uyaroğlu, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: Saglik Bilimleri University
Record Dates: First submitted 2021-03-08; First posted 2021-03-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: ICU Patients; ICU Acquired Weakness
Keywords: Physical Function; Critical İll; ICU Acquired Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation of the Chelsea Critical Care Physical Assesment Tools — The validation of the CPAX tools will focus on the validity of constructs, internal consistency reliability and test-retest reliability. PFIT used for criterion validity.

SUMMARY:
This study is aimed at providing an translation and cross-cultural adaptation of Chelsea Critical Care Physical Assesment Tool (CPAx) and tested its reliability and validity.

DETAILED DESCRIPTION:
Survival has increased in the ICU due to technological developments , but physical disability after discharge has become an important problem. İntensive Care Unit Acquired Weakness(ICU-AW) is seen in most of the patients admitted in this unit. The biggest reasons for ICU-AW are; sepsis, multiple organ failure and prolonged mechanical ventilation. The use of measurement tools to evaluate disabilities during stay and after discharge in intensive care unit, is a subject that has been researched all over the world.. These measurement tools provide; monitoring and evaluation during the ICU admission and assessment efficacy of treatment in the unit. The Chelsea Critical Care Physical Assessment Tool(CPAX) has been shown to valid, reliable and to exhibited strong clinimetric properties. CPAx is a numerical measurement tool, rated according to the 6-point Guttman Scale, from complete dependence to independence and consist of ten physical function parameters. This study is aimed at providing an translation and cross-cultural adaptation of Chelsea Critical Care Physical Assesment Tool (CPAx) and tested its reliability and validity. The protocol includes a pre-test of the Turkish version on 10 patients, a final revision, and a validation on a sample of 40 İCU patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Critical adult patients
* Patients who were hospitalized for more than 48 hours in an ICU

Exclusion Criteria:

* Unstable fracture
* Limb deformities and dysfunction
* Myasthenia gravis
* Neuromuscular dysfunction
* Patients who diagnosed COVİD-19

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Chelsea Critical Care Physical Assesment Tools | three days
  The Chelsea critical care physical assessment (CPAx) is a measurement tool used to assess physical function in the ICU. The Chelsea critical care physical assessment (CPAx) tool is an outcome measure designed to assess 10 domains of physical ability: respiratory function, cough, bed mobility, supine to sitting on the edge of the bed, dynamic sitting, sit to stand, standing balance, transferring from bed to chair, stepping and grip strength.
  The validation of the CPAX tools will focus on the validity of constructs, internal consistency reliability and test-retest reliability.

SECONDARY OUTCOMES:
Physical Function in Intensive Care Test | three days
  The PFIT is a test that measures function status of patients with a variety of conditions in the ICU. It includes 5 items: amount of assistance for sit-to-stand transfers, strength for shoulder flexion, strength for knee extension, marching in place, and an upper extremity endurance task of arm elevation to 90 degrees of shoulder flexion.
  PFIT used for criterion validity.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, Ass.Prof, Study Director — Saglik Bilimleri Universitesi; Mehmet Burak Uyaroğlu, PT, MSc, Principal Investigator — Saglik Bilimleri Universitesi; Sümeyye Akcay, PT, MSc, Study Chair — Saglik Bilimleri Universitesi; Gamze Koyutürk, PT, MSc, Study Chair — Saglik Bilimleri Universitesi; Hakan Parlak, MD, Study Chair — Istinye University Bahcesehir Hospital; Kürsat Baydilli, PhD, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Mehmet Burak Uyaroğlu, Istanbul, Turkey (Türkiye)